CLINICAL TRIAL: NCT04952740
Title: Application of Index of Microcirculatory Resistance to Evaluate Myocardial Protection After Ischemic Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013127
Record Dates: First submitted 2021-06-29; First posted 2021-07-07 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2014-01

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic postconditioning (Experimental): Routine PCI operations (including thrombus aspiration, stent injection, application of GPIIb/IIIa, etc.) + immediate post-ischemic adaptation: 30 seconds balloon inflation and 30 seconds deflation for 3 cycles
  Interventions: Procedure: IPC+PCI
- No Ischemic postconditioning (Active Comparator): Routine PCI operations (including thrombus aspiration, stent injection, application of GPIIb/IIIa, etc.)
  Interventions: Procedure: No IPC

INTERVENTIONS:
Procedure: IPC+PCI — Routine PCI operations (including thrombus aspiration, stent injection, application of GPIIb/IIIa, etc.) + immediate post-ischemic adaptation: 30 seconds balloon inflation and 30 seconds deflation for 3 cycles
  Other Names: Ischemic postconditioning
  Arms: Ischemic postconditioning
Procedure: No IPC — Routine PCI operations (including thrombus aspiration, stent injection, application of GPIIb/IIIa, etc.
  Other Names: Routine PCI
  Arms: No Ischemic postconditioning

SUMMARY:
To evaluate the protective effect of IPC on the myocardial microcirculation response through IMR and the predictive value of IMR on the degree of myocardial reperfusion and the prognosis of patients.

DETAILED DESCRIPTION:
This study is a clinical randomized controlled study, applying index of microcirculatory resistance (IMR) to evaluate the myocardial protection of ischemic postconditioning (IPC) in patients receiving direct PCI treatment for acute myocardial infarction.IMR is a quantitative evaluation index of microcirculation status. IPC has been reported to reduce ischemia-reperfusion injury and has a myocardial protective effect.The research plan divides patients into IPC and non-IPC groups at random. After the infarction-related artery is successfully implanted with a stent, the pressure guide wire is used to measure IMR and CFR in the state of maximal expansion of the microcirculation induced by intravenous ATP infusion.And analyze whether there are differences in indicators between the two groups and the relationship between these indicators and the patient's myocardial level reperfusion, cardiac function and prognosis.The purpose is to evaluate the myocardial protection of IPC and the predictive value of IMR on the degree of myocardial reperfusion and the prognosis of patients. It is expected that the target IPC can improve the IMR value, and IMR can predict the degree of myocardial reperfusion and cardiac function and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, no gender limit;
* First episode of STEMI (diagnostic criteria: ischemic chest pain lasting ≥30min; ST-segment elevation in two or more adjacent leads on the ECG or new left bundle branch block; with or without elevated myocardial markers), The onset time is within 12 hours, and emergency interventional treatment is planned;
* Agree and cooperate to participate in this research.

Exclusion Criteria:

* Old myocardial infarction;
* Killip grade of cardiac function ≥ grade III or cardiogenic shock;
* Systolic blood pressure ≤100mmHg;
* Bradycardia, HR<60pbm, or AVB above II degree;
* Past history of asthma or severe COPD;
* Severe liver and kidney dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
IMR | detected immediately after percutaneous coronary intervention
  index of microcirculatory resistance measured during coronary intervention.

SECONDARY OUTCOMES:
MACEs after PCI | 6 months
  MACEs includes cardiogenic death, non-fatal myocardial infarction, malignant arrhythmia, unplanned revascularization, unstable angina pectoris requiring hospitalization and severe heart failure requiring hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Lijun, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No